CLINICAL TRIAL: NCT06110845
Title: CLinical Evaluation Of a comPuter Algorithm To Report BreAst cAncers
Brief Title: CLinical Evaluation Of a comPuter Algorithm To Report BreAst cAncers (CLEOPATRAA)
Acronym: CLEOPATRAA
Status: Not yet recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other); 4DPath (Unknown)
Responsible Party: Sponsor
Other Study IDs: HP22/152913
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Digital Pathology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: QPlasia OncoReader Breast (QPORB) — Automated diagnostic algorithm

SUMMARY:
The goal of this non-interventionist observational study is to test the performance of a computer algorithm (QPORB) which examines breast cancer biopsy digital images to provide diagnostic support. The main question[s] it aims to answer are:

1. The principal research aim is to determine whether 4D Path's Technology Q-Plasia OncoReader Breast, that has been developed in the research setting, works robustly in the clinical environment (i.e. to define its real-life clinical utility) in terms of breast carcinoma grading and molecular subtyping
2. The secondary research aim is to perform an economic analysis alongside the trial in order to establish the time, resource and cost savings that the technology could afford the NHS, the ideal price point for engaging with the technology and the cost:benefit ratio for evaluation by the National Institute for Clinical Excellence
3. The tertiary research aim is to gather long-term follow-up data to better understand long-term response to therapy and prognosis and potential future uses of the algorithm

Participants's specimens will be tested alongside routine clinical workflows without intervention or consent. Researchers will compare the algorithm's results to those of routine diagnostic standard of care workflows.

DETAILED DESCRIPTION:
This study follows on from work conducted over the last 4 years focusing on developing computer-aided diagnostic algorithms in histopathology, with a focus on the detection and typing of breast cancer. The algorithm extracts information from the same digital image of a breast biopsy glass slide as used by pathologists to make a diagnosis. The algorithm can identify the presence of invasive cancer, grade it (i.e. how aggressive it looks) and determine its molecular subtype, all from the same image and in a single step. Whilst a pathologist can identify invasive cancer and grade it on a biopsy specimen, grading is inconsistent across reporting clinicians (i.e. prone to inter-observer variability) and only about 80% aligned with the 'true' grade of the tumour obtained at surgery. Moreover, additional time-consuming and expensive laboratory tests are required for molecular subtyping. They are however essential for informing oncologists of the most effective/targeted therapy for the patient in each case. The aim of this study is to perform a final real-life acid test of the technology in the clinical environment separately but in parallel with routine diagnostic services. If successful, the technology will have acquired a sufficient body of data to convince end-users and regulatory bodies of its merit and will effectively make it ready for deployment in the clinical environment. In that domain, this diagnostic solution health economics assessment will run alongside the clinical evaluation of the algorithm to analyse and compare cost and time-related factors between the routine clinical service and the algorithm workflow. This will provide further information required by regulatory bodies to aid the consideration of utilising the technology within current health systems. Furthermore, follow-up data will be collected at 5 and 10 years to investigate patient prognosis and treatment response as well as future potential applications of the technology.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a breast biopsy specimen processed at the pathology laboratory at SJUH, LTHT.

Exclusion Criteria:

* Age <16 or >110 years, non-carcinoma malignancies (e.g., sarcomas, malignant phyllodes tumours), carcinomas not arising from within the breast (e.g., cutaneous malignancies).

Ages: 16 Years to 110 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients biopsied for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2034-11-30 (Estimated)

PRIMARY OUTCOMES:
Concordance | 1 year
  The principal research aim is to determine whether 4D Path's Technology Q-Plasia OncoReader Breast, that has been developed in the research setting, works robustly in the clinical environment (i.e. to define its real-life clinical utility) in terms of breast carcinoma grading and molecular subtyping

SECONDARY OUTCOMES:
Health Economics evaluation | 6 months
  The secondary research aim is to perform an economic analysis alongside the trial in order to establish the time, resource and cost savings that the technology could afford the NHS, the ideal price point for engaging with the technology and the cost:benefit ratio for evaluation by the National Institute for Clinical Excellence

OTHER OUTCOMES:
Long term follow-up | 10 years
  The tertiary research aim is to gather long-term follow-up data to better understand long-term response to therapy and prognosis and potential future uses of the algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- St James's University Hospital, Leeds Teaching Hospitals Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not data shared with other researchers